CLINICAL TRIAL: NCT02406859
Title: Bowel Biofeedback Training to Improve Bowel Function in Individuals With SCI
Brief Title: Utility of an Animated Bowel Biofeedback Training Routine to Improve Bowel Function in Individuals With SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: B1915-P; KOR-13-010 (Other: James J. Peters Veterans Affairs Medical Center)
Record Dates: First submitted 2015-02-19; First posted 2015-04-02 (Estimated); Results first posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-08

CONDITIONS: Spinal Cord Injury; Constipation; Fecal Incontinence; Neurogenic Bowel
Keywords: Spinal Cord Injury; Constipation; Fecal Incontinence; Neurogenic Bowel; Bowel Biofeedback; Manometry
MeSH Terms: conditions — Spinal Cord Injuries; Constipation; Fecal Incontinence; Neurogenic Bowel

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anorectal Manometry (Experimental): Part 1 [Anorectal Manometry]: Fifty SCI subjects and 15 AB subjects will undergo anorectal manometry and a baseline assessment of level of constipation or frequency of fecal incontinence (FI). Additional 10 able-bodied subjects will be enrolled to serve as controls. The 10 Question Bowel Survey and Incontinence Scale will be administered.
  Interventions: Behavioral: Anorectal Manometry
- Bowel Biofeedback Training (Experimental): Part 2 [Bowel Biofeedback]: A subgroup of 20 subjects who participated in the first arm of the study (Anorectal Motility) and report either constipation or fecal incontinence will be asked to participate in 12 weeks of twice weekly, biofeedback training. The biofeedback training will consist of in-lab exercises that are paired with a visual feedback. Anorectal manometry and bowel surveys will be repeated after the training session to assess the effects of bowel biofeedback on anorectal function.
  Interventions: Behavioral: Bowel Biofeedback

INTERVENTIONS:
Behavioral: Bowel Biofeedback — Subjects will complete 2 sessions twice a week for 6 weeks of bowel biofeedback training. Subjects will be asked to squeeze and bear down for a period of 5 seconds followed by rest for 10seconds. Following the training, each subject will complete similar training at home for 6 weeks.
  Arms: Bowel Biofeedback Training
Behavioral: Anorectal Manometry — Subjects will undergo an anorectal manometry to establish baseline pressure characteristics. If subjects qualify for biofeedback training, they will complete two additional manometries to track the changes occuring during training.
  Arms: Anorectal Manometry

SUMMARY:
An injury to the spinal cord results in a number of secondary medical problems, including the inability to voluntarily control the bowels. Depending on the severity and location of the injury, remaining bowel function differs, and can include any combination of the following: constipation (prolonged stool retention), difficulty with evacuation (difficultly moving bowels), fecal incontinence (problems retaining stool until it is appropriate to move the bowels). Most of the current medications and treatment options address problems of constipation and difficulty with evacuation, but there are few options for individuals who suffer from incontinency. In this study, the investigators propose to study, in detail, anorectal muscle function in individuals with spinal injury - the investigators will do so using new technology called high resolution manometry - which will present the investigator with a 3 dimensional representation of the pressure profile of the anorectal muscles as the subject attempts different maneuvers. A subgroup with representatives of all levels and completeness of injury and anorectal muscle function will be enrolled to participate in six weeks of biofeedback training to see if their bowel function can be improved. During these six weeks, the subjects will be asked to visit the laboratory twice a week in order to be trained by the research team on how to improve their anorectal strength and function in response to visual cues. After the six weeks, another manometry study will be performed. Subjects will then be sent home and asked to perform a series of home exercises for another 6 weeks, after which they will asked to return for a third and final manometry study.

DETAILED DESCRIPTION:
Neurogenic bowel characteristics differ among spinal cord injured (SCI) individuals, and appear to depend primarily on the level and completeness of injury. It is thought that upper motor neuron lesions in the spinal cord above L1-2 results in a hyperreflexive bowel with increased colonic wall tone and loss of cortical control over the relaxation of the external anal sphincter (EAS). These changes result in chronic high sphincter tone and dyssynergic defecation. The main symptoms in these patients are constipation and fecal retention, or difficulty with evacuation (DWE). In many of these individuals, some nerve connections between the spinal cord and the colon may be preserved, and stool propulsion and reflex coordination may remain intact and under control of the central nervous system. Furthermore, individuals with spinal lesions above T7 experience loss of voluntary control over abdominal muscles and an inability to increase intra-abdominal pressure, which results in more DWE and constipation. Lower motor neuron (LMN) lesions in the spinal cord below L1-2 result in the interruption of the centrally mediated innervation to the bowel, which causes slowing of peristalsis, a flaccid EAS, and atonic levator ani muscles. This is also called an areflexic bowel. The main symptoms in these patients are constipation from slowed peristalsis and fecal incontinence (FI) from atonic EAS and levator ani muscles. While the symptoms of bowel dysfunction in persons with SCI are known, function and motility of the anal canal have not been documented in this population. Anorectal manometry can provide valuable information about sphincter strength, defecation dynamics and reflex mechanisms. New high-resolution anorectal manometric systems (Given Imaging, Duluth, GA), simultaneously captures pressure data from the rectum, IAS, EAS and atmosphere. High resolution manometry also allows for much clearer display of pressure events compared to line tracing series, and direction of contractions are much easier to discern. To date, anorectal high resolution topographical studies have not been conducted in a SCI population.

Modalities in which the patient can be trained to control the internal anal sphincter (IAS) and EAS are promising solutions to FI, and have been shown to be useful in able bodied (AB) populations. For example, anorectal biofeedback methods teach patients to recognize sensations of a distended rectum while also teaching abdominal or pelvic muscles to voluntarily contract for short periods of time in order to improve continence. Such biofeedback modalities have also been shown to decrease constipation in AB populations by teaching proper external sphincter relaxation and rectal muscle contraction. The concept of biofeedback is based on principles of operant conditioning, in which information concerning a normally subconscious physiological function in relayed to patients and that become actively engaged in learning to consciously control this function. During bowel (re)training programs, patients are provided with visual feedback on voluntary and reflex sphincter and rectal muscle contractions, so that they can learn to recognize diffuse sensations and gradually regain control.

ELIGIBILITY:
Inclusion Criteria:

* Chronic SCI (duration over 1 year)
* Able-bodied (no SCI)

Exclusion Criteria:

* Contraindication to bowel biofeedback
* Currently pregnant or trying to become pregnant
* Inability to provide informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Korsten, MD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aloysius MM, Korsten MA, Radulovic M, Singh K, Lyons BL, Cummings T, Hobson J, Kahal S, Spungen AM, Bauman WA. Lack of improvement in anorectal manometry parameters after implementation of a pelvic floor/anal sphincter biofeedback in persons with motor-incomplete spinal cord injury. Neurogastroenterol Motil. 2023 Nov;35(11):e14667. doi: 10.1111/nmo.14667. Epub 2023 Sep 25. PMID 37743783

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: American Spinal Cord Injury Association (ASIA) exams were administered to all subjects with spinal cord injury to determine severity of injury and whether the participant meets the criteria to participate in bowel biofeedback training portion.
Groups:
- Able Body Participants: Anorectal Manometry: Able bodied subjects will undergo anorectal manometry and a baseline assessment of level of constipation or frequency of fecal incontinence (FI). Subjects will undergo an anorectal manometry to establish baseline pressure characteristics.
- Complete Spinal Cord Injury (ASIA A): Anorectal Manometry: Subjects with ASIA A spinal cord injury will undergo anorectal manometry and a baseline assessment of level of constipation or frequency of fecal incontinence (FI). The 10 Question Bowel Survey and Incontinence Scale will be administered. Subjects will undergo an anorectal manometry to establish baseline pressure characteristics.
- Incomplete Spinal Cord Injury (ASIA B,C,D): Part 1 Anorectal Manometry and 10 Question Bowel Survey
  Part 2 [Bowel Biofeedback]: A subgroup of subjects who participated in the first arm of the study (Anorectal Motility) and report either constipation or fecal incontinence will be asked to participate in 12 weeks of twice weekly, biofeedback training. The biofeedback training will consist of in-lab exercises that are paired with a visual feedback. Anorectal manometry and bowel surveys will be repeated after the training session to assess the effects of bowel biofeedback on anorectal function.
  Bowel Biofeedback: Subjects will complete 2 sessions twice a week for 6 weeks of bowel biofeedback training. Subjects will be asked to squeeze and bear down for a period of 5 seconds followed by rest for 10seconds. Following the training, each subject will complete similar training at home for 6 weeks.
Period: Part 1 - Manometric Parameters
Arm/Group | Able Body Participants | Complete Spinal Cord Injury (ASIA A) | Incomplete Spinal Cord Injury (ASIA B,C,D)
Started | 15 | 14 | 21
Completed | 12 | 13 | 17
Not Completed | 3 | 1 | 4
Period: Part 2 - Biofeedback Training
Arm/Group | Able Body Participants | Complete Spinal Cord Injury (ASIA A) | Incomplete Spinal Cord Injury (ASIA B,C,D)
Started | 12 | 13 | 17
Completed | 12 | 13 | 17
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The information available was collected from participants that participated in in part 1 of the study as opposed to those participants that consented to the study. The subjects that consented but did not start part 1 are not included in this information.
Groups:
- Able Bodied Participants: The representation of this group are those participants with no known spinal cord injury and full motor function.
- Complete Spinal Cord Injury (ASIA A): The representation of this group are those participants with known spinal cord injury and medically diagnosed with an American spinal cord injury rating of A. This exam will delineate that the individual has a complete lack of motor and sensory function below the level of injury.
- Incomplete Spinal Cord Injury (ASIA B, C, D): The representation of this group are those participants with known spinal cord injury and medically diagnosed with an American spinal cord injury rating of B,C or D. This exam will delineate that the individual falls within the range of having some sensation below the level of injury to most motor function and sensation being preserved below the level of injury.
- Total: Total of all reporting groups
Arm/Group | Able Bodied Participants | Complete Spinal Cord Injury (ASIA A) | Incomplete Spinal Cord Injury (ASIA B, C, D) | Total
Number analyzed (Participants) | 12 | 13 | 17 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 14 | 37
  >=65 years | 0 | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 2
  Male | 12 | 13 | 15 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  United States | 12 | 13 | 17 | 42
Mean Sphincteric Pressure (mm Hg) [Mean (Standard Deviation); unit: mmHg] — Measured by high resolution anorectal manometry
  mmHg | 77.9 (21.9) | 67.1 (31.8) | 65.2 (21.4) | 72.0 (26.2)

OUTCOME MEASURES:

1. Primary Outcome: Baseline Motility (Anorectal Sensation and Strength) Characteristics
Description: We aim to assess the following baseline motility characteristics: maximum sphincter pressure (resting and squeezing pressure), mean sphincter pressure, residual anal and intrarectal pressure (high pressure zone), and recto-anal pressure differential (difference of intrarectal and residual anal pressures) in persons with chronic spinal cord injury (SCI) and able bodied (AB) subjects.
Time Frame: 1 Session (Baseline Anorectal Manometry Assessment)
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Able Bodied Participants: Part 1 [Anorectal Manometry]: Able bodied subjects will undergo an anorectal manometry to establish baseline pressure characteristics to serve as a comparison group for the SCI complete and incomplete baseline groups.
- Complete Spinal Cord Injury (ASIA A): Part 1 [Anorectal Manometry]: Subjects with complete spinal cord injury will undergo an anorectal manometry to establish baseline pressure characteristics, to compare with the incomplete spinal cord injury group.
- Incomplete Spinal Cord Injury (ASIA B, C, D): Part 1 [Anorectal Manometry]: Subjects with incomplete spinal cord injury will undergo an anorectal manometry to establish baseline pressure characteristics. If subjects qualify for biofeedback training, they will complete two additional manometries to track the changes occurring due to training.
Arm/Group | Able Bodied Participants | Complete Spinal Cord Injury (ASIA A) | Incomplete Spinal Cord Injury (ASIA B, C, D)
Number analyzed (Participants) | 12 | 12 | 20
mmHg
  Intra-rectal Pressure | 105 (35) | 34.4 (29) | 30 (19)
  Mean Sphincter Pressure | 77.9 (21.9) | 67.1 (31.8) | 65.2 (21.4)
  Max Sphincter Pressure | 253 (101) | 81.1 (12.3) | 108.9 (64)
  Residual anal Pressure | 169.3 (55) | 61.4 (42) | 73.8 (30)
  Recto-anal Pressure Differential | -63 (31) | -27 (7) | -44 (20)

2. Secondary Outcome: Change in Rectal and Sphincter Pressure Due to Bowel Biofeedback Training in Individuals With Incomplete SCI.
Description: Changes in maximum rectal and sphincter pressures generated during "squeeze" and "bear down" maneuvers performed during anorectal manometric studies pre-biofeedback training (baseline) and post-guided (part 1) and self-guided (part 2) biofeedback training.
Time Frame: Baseline, post- 6 week guided biofeedback training (weeks 1-6), post- 6 week self-guided biofeedback training (weeks 7-12).
Population: Participants with Incomplete Spinal Cord Injury (ASIA B, C, D). 17 participants with SCI (incomplete) completed baseline procedures; of those 17, 13 participants completed bowel biofeedback training part 1 (guided) and part 2 (self-guided).
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Incomplete Spinal Cord Injury (ASIA B, C, D); Baseline (Pre-bowel Biofeedback Training): Baseline characteristics were assessed. Squeezing and bearing down maneuvers were attempted.
- Incomplete Spinal Cord Injury (ASIA B, C, D); Bowel Biofeedback Training Part 1 (Guided): Bowel Biofeedback Training (Guided): Subjects will complete 2 sessions twice a week for 6 weeks of bowel biofeedback training. Subjects will be asked to squeeze and bear down for a period of 5 seconds followed by rest for 10 seconds.
- Incomplete Spinal Cord Injury (ASIA B, C, D); Bowel Biofeedback Training Part 2 (Self Guided): Bowel Biofeedback Training (Self Guided): Subjects will complete an at home training program 2 times a week over a 6 week period.
Arm/Group | Incomplete Spinal Cord Injury (ASIA B, C, D); Baseline (Pre-bowel Biofeedback Training) | Incomplete Spinal Cord Injury (ASIA B, C, D); Bowel Biofeedback Training Part 1 (Guided) | Incomplete Spinal Cord Injury (ASIA B, C, D); Bowel Biofeedback Training Part 2 (Self Guided)
Number analyzed (Participants) | 17 | 13 | 13
mmHg
  Max Sphincter Pressure | 71.39 (24.32) | 61.21 (23.36) | 61.41 (20.60)
  Mean Sphincter Pressure | 65.23 (21.49) | 55.58 (21.29) | 56.05 (19.69)
  Squeeze Max Pressure | 109.54 (63.57) | 105.96 (63.20) | 106.69 (52.06)
  Residual Anal Pressure | 73.79 (30.38) | 80.09 (34.36) | 84.35 (32.83)
  Intrarectal Pressure | 29.75 (19.98) | 38.53 (30.17) | 37.48 (37.52)

3. Secondary Outcome: Changes in Recto-anal Inhibitory Reflex (RAIR) Due to Bowel Biofeedback Training in Individuals With Incomplete SCI.
Description: Changes to the sensitivity and strength of response of the recto-anal inhibitory reflex (RAIR) in response to rectal distension.
  Outcome measure clarification: Minimal balloon volume, in cc, which was the threshold at which anorectal sensation was perceived by subjects with incomplete SCI, as assessed through High Resolution Manometry (HRM)
Time Frame: as for outcome 2
Population: Subjects that reached the maximum set limit of balloon inflation with no sensation were set as a non-recordable value.
Measure: Mean (Standard Deviation); unit: cc
Groups:
- Incomplete Spinal Cord Injury (ASIA B, C, D); Baseline (Pre-bowel Biofeedback Training): Subjects with incomplete spinal cord injury were asked to complete a balloon distension test pre-biofeedback training (baseline). The rectal balloon was distended until an urge to defecate occurs or to a maximum of 150 CCs.
- Incomplete Spinal Cord Injury (ASIA B, C, D); Bowel Biofeedback Training Part 1 (Guided): Bowel Biofeedback Training (Guided): Subjects with Incomplete SCI were asked to perform a balloon distention test following six week of guided bowel biofeedback training.
- Incomplete Spinal Cord Injury (ASIA B, C, D); Bowel Biofeedback Training Part 2 (Self Guided): Bowel Biofeedback Training (Self Guided): Subjects with Incomplete SCI were asked to perform a balloon distention test following 6 weeks of self-guided bowel biofeedback training.
Arm/Group | Incomplete Spinal Cord Injury (ASIA B, C, D); Baseline (Pre-bowel Biofeedback Training) | Incomplete Spinal Cord Injury (ASIA B, C, D); Bowel Biofeedback Training Part 1 (Guided) | Incomplete Spinal Cord Injury (ASIA B, C, D); Bowel Biofeedback Training Part 2 (Self Guided)
Number analyzed (Participants) | 17 | 13 | 13
cc
  Balloon Volume - First Sensation | 41.87 (17.21) | 35.00 (14.46) | 51.82 (30.27)
  Balloon Volume - Urge to Defecate | 63.13 (30.92) | 59.17 (25.39) | 67.00 (29.83)

4. Secondary Outcome: Change in Subjective Bowel Care Due to Guided and Self-Guided Biofeedback Training in Individuals With Incomplete SCI
Description: Constipation and fecal Incontinence was assessed in participants with incomplete SCI by the Ten Question Bowel Survey. This survey is based on a scale 1-5; a lower score represents fewer bowel management difficulties (better functioning). Survey was administered at baseline (pre-training), and post- guided (part 1) and self-guided (part 2) bowel biofeedback training.
Time Frame: as for outcome 2
Population: Subjects with Incomplete SCI, pre (baseline) and post guided and self-guided biofeedback training.
Measure: Mean (Standard Deviation); unit: Score on scale
Groups:
- Incomplete Spinal Cord Injury (ASIA B, C, D); Baseline (Pre-bowel Biofeedback Training): Baseline - subjects with incomplete Spinal Cord Injury (ASIA B, C, D) were asked to complete the 10 Question Bowel Survey (QBS) prior to biofeedback training.
- Incomplete Spinal Cord Injury (ASIA B, C, D); Bowel Biofeedback Training Part 1 (Guided): Bowel Biofeedback Training (Guided): Subjects with incomplete Spinal Cord Injury (ASIA B, C, D) were asked to complete the 10 QBS following 2 sessions twice a week for 6 weeks of bowel biofeedback training.
- Incomplete Spinal Cord Injury (ASIA B, C, D); Bowel Biofeedback Training Part 2 (Self Guided): Bowel Biofeedback Training (Self Guided): Subjects with incomplete Spinal Cord Injury (ASIA B, C, D) were asked to complete the 10 QBS following an at home training program 2 times a week over a 6 week period..
Arm/Group | Incomplete Spinal Cord Injury (ASIA B, C, D); Baseline (Pre-bowel Biofeedback Training) | Incomplete Spinal Cord Injury (ASIA B, C, D); Bowel Biofeedback Training Part 1 (Guided) | Incomplete Spinal Cord Injury (ASIA B, C, D); Bowel Biofeedback Training Part 2 (Self Guided)
Number analyzed (Participants) | 15 | 13 | 13
Score on scale
  Frequency of Bowel Movement Scale:10Question Bowel Survey (QBS) Range:1 (≥7 times/week) to 5(None) | 2.53 (1.25) | 2.54 (.97) | 2.38 (1.33)
  Bowel Evacuation Time: Scale: 10 QBS Range: 1 (5-15min/day) to 5 (≥3hrs/day) | 2.20 (1.32) | 1.69 (1.03) | 2.00 (1.15)
  Leakage (per week): Range: 1 (leakage 0 times) to 5 (leakage ≥7 times) | 1.13 (.35) | 1.23 (.44) | 1.31 (.48)
  Enemas (per week): Range: 1 (none used) to 5 (used every time) | 2.13 (1.64) | 2.08 (1.71) | 2.23 (1.79)
  Oral Medications (per week): Range: 1 (none used) to 5 (used every time) | 2.33 (1.84) | 2.00 (1.73) | 2.54 (2.03)
  Digital Stimulation (per week): Range: 1 (none) to 5 (every time) | 1.80 (1.42) | 1.69 (1.49) | 2.38 (1.85)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the entirety of the study which lasted approximately 12 weeks for each subject.
Groups:
- Able Body Participants: Anorectal Manometry: Able bodied subjects underwent anorectal manometry as a baseline assessment. Anorectal manometry is the only procedure that put this group an greater than no risk.
- Complete Spinal Cord Injury (ASIA A): Anorectal Manometry: SCI subjects medical designated with an injury severity score of ASIA A underwent anorectal manometry as a baseline assessment. Anorectal manometry is the only procedure that put this group an greater than no risk.
- Incomplete Spinal Cord Injury (ASIA B,C,D): Anorectal Manometry: SCI subjects medical designated with an injury severity score of ASIA B,C and D underwent anorectal manometry as a baseline assessment. Participants were then asked to participate in 12 weeks of twice weekly, biofeedback training. The biofeedback training will consist of in-lab exercises that are paired with a visual feedback. Anorectal manometry was repeated after the training session to assess the effects of bowel biofeedback on anorectal function.
Arm/Group | Able Body Participants | Complete Spinal Cord Injury (ASIA A) | Incomplete Spinal Cord Injury (ASIA B,C,D)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/21
Other Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/21

LIMITATIONS AND CAVEATS:
The trial was limited by a small number of participants due to strict inclusion and exclusion criteria

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/59/NCT02406859/Prot_000.pdf
  • Statistical Analysis Plan (2013-03-10): https://cdn.clinicaltrials.gov/large-docs/59/NCT02406859/SAP_001.pdf
  • Informed Consent Form (2016-09-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT02406859/ICF_002.pdf